CLINICAL TRIAL: NCT06076265
Title: Quantitative Detection of CEA mRNA in the Smog and Tissue Exudate Whole Process Collected During Laparoscopic (Robotic) Radical Gastrectomy in Gastric Cancer Patients: Study Protocol for a Single Center Prospective, Single-arm, Longitudinal Pilot Study（SMOG 01Study）
Brief Title: Quantitative Detection of CEA mRNA in the Smog and Tissue Exudate Whole Process Collected During Laparoscopic (Robotic) Radical Gastrectomy in Gastric Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: SMOG01
Record Dates: First submitted 2023-09-20; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer
Keywords: Advanced Gastric Cancer; Laparoscopic(Robotic) Gastrectomy; RT-PCR; CEA; Free intraperitoneal tumor cells
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm group
  Interventions: Procedure: Radical Gastric Cancer Surgery

INTERVENTIONS:
Procedure: Radical Gastric Cancer Surgery — Laparoscopic (robotic) radical surgery for gastric cancer

SUMMARY:
The purpose of this SMOG 01 study is to observe the possibility of intraperitoneal dissemination of tumor cells throughout the entire laparoscopic (robotic) radical gastrectomy for gastric cancer and explore its related mechanisms and potential clinical significance with peritoneal metastasis.

DETAILED DESCRIPTION:
Cytological examination of peritoneal lavage fluid has become an important parameter for pathological staging and prognosis judgment of gastric cancer. However, the vast majority of previous studies have only focused on collecting peritoneal lavage fluid through laparotomy or laparoscopic exploration for cytological and tumor marker monitoring as further tumor staging. Unfortunately, there is no research focusing on whether laparoscopic (or robotic) surgery under the carbon dioxide pneumoperitoneum environment can cause the iatrogenic spread of cancer cells, and there is also a lack of a practical and feasible method to collect smog and tissue exudates generated throughout the entire surgical process for cytological monitoring, to determine whether laparoscopic surgery itself may cause the iatrogenic spread of tumor cell, to uncover the potential mechanisms and propose appropriate preventive measures of peritoneal metastasis. Therefore, the investigators have designed a special device to collect smog and tissue exudates generated during laparoscopic or robotic radical gastrectomy to determine whether there is a possibility of iatrogenic cancer cell dissemination in the abdominal cavity throughout the entire course of laparoscopic or robotic surgery by using RT-PCR to detect CEA mRNA, which can become one of the reasons for gastric cancer peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Gastric adenocarcinoma confirmed by preoperative pathology
* Endoscopic and CT/MRI enhanced examination confirmed that cT1-4aN0-3M0 has the possibility of resection
* To undergo radical gastrectomy (laparoscopic or robotic) under general anesthesia+/- epidural anesthesia (carbon dioxide pneumoperitoneum)
* Willing and able to comply with the research protocol
* Reach a written consent agreement before registration, and fully realize the right to withdraw from the study at any time without any loss

Exclusion Criteria:

* Urgent surgery is required due to tumor emergencies (such as bleeding, perforation, and obstruction)
* Extensive peritoneal metastasis can be seen during intraoperative exploration
* Other diseases requiring simultaneous surgery
* Patients with ascites
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients over 18 years old who plan to undergo radical gastrectomy for gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Positive detection rate of CEA | Supervision of the whole operation: collection of peritoneal lavage fluid at three time points, before the start of the operation, during the operation, and at the end of the operation
  Positive detection rate of CEA

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Yanbing, MD, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR